CLINICAL TRIAL: NCT05485506
Title: Effects of a Multimodal Exercise Program on the Kinematics and Sprint Performance of Young Rugby Players: an Experimental Study.
Brief Title: Multimodal Exercises on Sprint Performance of Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 278CER22
Record Dates: First submitted 2022-07-30; First posted 2022-08-03 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2022-07

CONDITIONS: Exercise Training; Rugby; Adolescent
Keywords: sprint performance; strength training; sprint kinematics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will add to their training routine a multimodal exercise program (two days per week, during six weeks). This program will include running technical drills, exercises for lumbopelvic stabilization and resisted sprints by using sled.
  Interventions: Other: Multimodal exercise program
- Control group (No Intervention): Control group will maintain their training routine.

INTERVENTIONS:
Other: Multimodal exercise program — Running technical drills: pogo, askip, dribble, scissor, etc. Exercises for lumbopelvic stabilization: mobility exercises, hip thrust, dead lift, lunge to skip.
  Resisted sprints by using a sled: resistance leading to a 60% and 30% of optimal load (previously calculated)
  Arms: Intervention group

SUMMARY:
This study is designed to evaluate the effects of a multimodal exercise program in the sprint performance and kinematics of adolescent rugby players. For this, an experimental study with an intervention group (IG) and a control group (CG) is designed. During 6 weeks of the 2022-2023 preseason of rugby seven, IG will include a multimodal exercise program in their training routine. Meanwhile, CG will maintain their training routine. The study will be developed in the Sport High Performance Centre of Balearic Islands during the season of rugby seven (from August to September, 2022). All rugby athletes from under-16 and under-18 autonomic rugby teams will be invited to participate in this study throughout an email invitation from their regional rugby federation. Prior to the beginning of the study, all participants will sign the inform consent, or their legal tutors in case of minors. The Ethical Committee of the local university approved this study (278CER22) according to the Declaration of Helsinki.

One week before intervention period, sociodemographic and sportive data will be registered (age, sex, body mass, height, and sport experience). Body mass and height will be evaluated with a ±100-g precision digital weight scale (Tefal, France) and a t201-t4 adult height scale (Asimed, Spain), respectively. Also, the rugby players will complete a familiarization process consisting on a standardized warm up and 3 progressive sprints (i.e. 30 m at 50%, 70% and 90% of maximal effort).

All testing procedure (pre-test and post-test) will be completed at a similar daytime (between 17h and 19h) on the same natural grass field. The test procedure listed in our study will consist on two maximal 30-m sprints to obtain mechanical variables of horizontal force-velocity profile and kinematics during sprinting.

Players from IG will perform a multimodal exercise program two days per week during six weeks. This program will include running technical drills, exercises for lumbopelvic stabilization and resisted sprints. This program will be supervised by two experts in this field.

The investigators hypothesize that those rugby players who add the multimodal exercise program to their training routine will increase mechanical and kinematics variables of sprint performance.

ELIGIBILITY:
Inclusion Criteria:

* to have at least 14 years old
* to have at least 2 years of experience as rugby player

Exclusion Criteria:

* to have sustained a lower limb or lumbopelvic injury during the previous 6 months to start of the study
* to have sustained a lower limb or spine surgery during the previous 12 months to start of the study

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Sprint performance | Change from baseline and between group differences in sprint performance after the intervention period of 6 weeks
  Sprint performance measured with MySprint. Resulting from maximal 30-m sprint, six pairs of brands with parallax corrected will be placed at 0, 5, 10, 15, 20 and 30 m to measure the five different split times in seconds during the 30-m trials. The camera, which records 240 frame per second, will be situated on a tripod (in the sagittal plane) 10 meters away from the fourth marker in meter 15.
Force-Velocity Profile (F-V) | Change from baseline and between group differences in horizontal force-velocity profile after the intervention period of 6 weeks
  F-V Profile measured by My Sprint App, resulting from maximal 30-m sprint, theorical maximal horizontal force (F0), maximal mechanical power output in the horizontal direction (Pmax), rate of decrease in RF with increasing speed during sprint acceleration (DRF), Slope of the linear F-V relationship (Sfv), Ratio of force (RF) and maximal value of RF (RFmax). The camera, which records 240 frame per second, will be situated on a tripod (in the sagittal plane) 10 meters away from the fourth marker in meter 15.
Sprint spatiotemporal and kinematics | Change from baseline and between groups in sprint spatiotemporal and kinematics at 6 weeks
  Sprint spatiotemporal and kinematics will be analyzed with Kinovea program (v.0.8.15). The following variables will be analyzed: contact time (s), length step (m; horizontal displacement between the toe tips at adjacent touchdowns), step rate (Hz; the reciprocal of step duration). Moreover, in the frame that the foot touchdown and the frame that the foot touch off trunk and hip (ipsilateral and contralateral) angles will be quantified. The camera, which records 240 frame per second, will be situated 9 meters away from 22.5 m on a tripod at a height of 1.1 meters in the sagittal plane.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero Franco, PhD, Study Director — University of the Balearic Islands
Locations (1):
- Sport High Performance Centre of Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayala F, Lopez-Valenciano A, Gamez Martin JA, De Ste Croix M, Vera-Garcia FJ, Garcia-Vaquero MDP, Ruiz-Perez I, Myer GD. A Preventive Model for Hamstring Injuries in Professional Soccer: Learning Algorithms. Int J Sports Med. 2019 May;40(5):344-353. doi: 10.1055/a-0826-1955. Epub 2019 Mar 14. PMID 30873572
- [Background] Brooks JH, Fuller CW, Kemp SP, Reddin DB. Incidence, risk, and prevention of hamstring muscle injuries in professional rugby union. Am J Sports Med. 2006 Aug;34(8):1297-306. doi: 10.1177/0363546505286022. Epub 2006 Feb 21. PMID 16493170
- [Background] Mendiguchia J, Castano-Zambudio A, Jimenez-Reyes P, Morin JB, Edouard P, Conceicao F, Tawiah-Dodoo J, Colyer SL. Can We Modify Maximal Speed Running Posture? Implications for Performance and Hamstring Injury Management. Int J Sports Physiol Perform. 2022 Mar 1;17(3):374-383. doi: 10.1123/ijspp.2021-0107. Epub 2021 Nov 18. PMID 34794121
- [Background] Mendiguchia J, Edouard P, Samozino P, Brughelli M, Cross M, Ross A, Gill N, Morin JB. Field monitoring of sprinting power-force-velocity profile before, during and after hamstring injury: two case reports. J Sports Sci. 2016;34(6):535-41. doi: 10.1080/02640414.2015.1122207. Epub 2015 Dec 9. PMID 26648237
- [Background] Mendiguchia J, Martinez-Ruiz E, Edouard P, Morin JB, Martinez-Martinez F, Idoate F, Mendez-Villanueva A. A Multifactorial, Criteria-based Progressive Algorithm for Hamstring Injury Treatment. Med Sci Sports Exerc. 2017 Jul;49(7):1482-1492. doi: 10.1249/MSS.0000000000001241. PMID 28277402
- [Background] Setuain I, Lecumberri P, Izquierdo M. Sprint mechanics return to competition follow-up after hamstring injury on a professional soccer player: A case study with an inertial sensor unit based methodological approach. J Biomech. 2017 Oct 3;63:186-191. doi: 10.1016/j.jbiomech.2017.08.010. Epub 2017 Aug 20. PMID 28844725
- [Background] Lahti J, Huuhka T, Romero V, Bezodis I, Morin JB, Hakkinen K. Changes in sprint performance and sagittal plane kinematics after heavy resisted sprint training in professional soccer players. PeerJ. 2020 Dec 15;8:e10507. doi: 10.7717/peerj.10507. eCollection 2020. PMID 33362970
- [Result] Sastre-Munar A, Jimenez-Reyes P, Romero-Franco N. Effects of a six-week multimodal training programme on the sprinting ability of adolescent rugby sevens players. J Sports Sci. 2023 Jun;41(10):990-998. doi: 10.1080/02640414.2023.2257514. Epub 2023 Sep 15. PMID 37712360